CLINICAL TRIAL: NCT04309630
Title: Comparison of Continuous Erector Spina Plan Block With Intercostal Block in Acute and Chronic Pain Control After Thoracotomy
Brief Title: Comparison of Continuous Erector Spina Plane Block With Intercostal Block in Acute and Chronic Pain Control After Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, ASS. PROFFESSOR, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-92-20
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intercostal block (Active Comparator): patients received intercostal block will be evaluated by visual analog score for pain assesment
  Interventions: Procedure: intercostal block
- erector spina plane block (Experimental): patients received erector spina plane block will be evaluated by visual analog score for pain assesment
  Interventions: Procedure: erector spina plane block

INTERVENTIONS:
Procedure: intercostal block — pain control by intercostal block
  Arms: intercostal block
Procedure: erector spina plane block — pain control by erector spina plane block
  Arms: erector spina plane block

SUMMARY:
Thoracotomy is associated with severe postoperative pain due to surgical incision, rib retraction or resection, and intercostal nerve damage. Pain management after thoracic surgery is extremely important for various reasons, including respiratory mechanics, decreased atelectasis, early mobilization, decreased opioid consumption, decreased hospital stay, and patient satisfaction.

Thoracic epidural analgesia and thoracic paravertebral blocks, although it comes to mind in the first place for thoracic surgery, the difficulty / failure of the application technique and the use of side effects such as spinal cord injury, pneumothorax and hypotension.

Alternative regional methods have come to the fore in recent years. Erector spina plan block (ESPB) is a recently defined interfacial plan block used for the treatment of thoracic neuropathic pain, trauma and acute pain after surgery.

Local anesthetic injection for ESPB can be applied both to the surface and deep into the erector spina muscle. When local anesthetic is applied deep into the erectral spina muscle, it has been demonstrated by the cadaver findings that the thoracic spinal nerves reach both the dorsal and ventral ramus with the spread of the paravertebral and intercostal areas. The thoracolumbar extension of the erector spina muscle allows wide cranio-caudal spread of injections in this plane and analgesia involving multiple dermatomes. This multisegmental analgesia allows ESPB to be used in pain management after thoracic or abdominal surgery.

Accompanied by ultrasound, ESPB is simple and reliable. With the easy recognition of sonoanatomy, the risk of damage to the surrounding tissues is negligible . If necessary, a permanent catheter can be placed that can be used to prolong analgesia time and can be used for both intraoperative and postoperative analgesia with catheter-mediated ESPB.

DETAILED DESCRIPTION:
After the approval of the ethics committee, patients with ASA I-II, elective thoracotomy plan will be informed that they will be included in the study before the operation and informed consent will be obtained. Routine preoperative anesthesia examinations of the patients will be performed. When patients come to the operating table, after routine monitoring of ECG, non-invasive blood pressure, pulse oximeter, BIS and TOF, sedation will be applied to patients.

After preoxygenation is performed with oxygen flow of 4 l / min, anesthesia induction will be applied to patients with propofol 3mg / kg and rocuronium 0.6mg / kg, and the patient will be intubated after sufficient muscle relaxation is achieved. Maintenance of anesthesia will be provided with BIS 40-60 with desflurane and 50% air + 50% O2. During the operation period, patients will receive 50mcg of fentanyl per hour for intraoperative analgesia and 10mg rocuronium to maintain muscle relaxation. At the end of the surgery, patients will be administered IV 1gr paracetamol and 4mg ondansetron to reduce the risk of vomiting postoperative nausea.

At the end of the surgery, thoracic vertebral spinous processes will be displayed by placing the linear ultrasound probe in the middle line at the level of T5 vertebra under the aseptic conditions while in the lateral decubitus position. Then, the transducer process of the subcutaneous adipose tissue, m.trapezius, m.rhomboideus major, m.erector spina and T5 vertebra will be displayed by shifting the probe 2-3cm laterally. After the needle placement is confirmed by hydrodissection with 3ml of 0.9% NaCl under the erector spina muscle, after 20ml 0.5% bupivacaine injection, the catheter will be placed in the 2-3cm intercostal area and the infusion of 2-4ml / hour 0.5% bupivacaine, daily total dose 400mg will not be exceeded. In the second group of patients, catheter will be placed in the intercostal area by the surgical team at the end of the surgery and 2-4ml / hour 0.5% bupivacaine infusion will be adjusted so that the total daily dose does not exceed 400mg.

After the anesthetic agent is terminated, when the TOF is 4, the effect of the muscle relaxant will be reversed by applying neostigmine and atropine to the patients. In order to provide analgesia to the patients in the postoperative period, the IV patient controlled analgesia device will be prepared as bolus with a 10-minute lock time, with the total dose of fentanyl not exceeding 1mcg / kg per hour, and will be started by explaining to the patients in the post-surgery department. If VAS> 4 and PCA bolus is insufficient, patients will receive paracetamol 1gr IV infusion.

Surgical procedures, incision length, operation time, total muscle relaxant and fentanyl doses used in the intraoperative period, the amount of fluid given to the patients, the amount of urine of the patients, the amount of bleeding during the operation, and the patient's blood pressure, heart rate and additional drug use will be recorded in the operation room.

Visual analogue scale (VAS) scores, satisfaction, nausea, vomiting, antiemetic use, itching complaints, mean artery at 30 minutes, 6,12,24,48,72 hours and postoperative time of chest withdrawal time. pressure, heart rate and saturation are monitored, the quality of the recovery will be evaluated with ALDRETE scoring and additional analgesic needs will be questioned. Patient controlled analgesia device will be requested at 30 minutes, 6, 12, 24 and 48 hours, and the number of bolus requested by the patient, the number of bolus delivered to the patient and the amount of drug will be recorded.

In the postoperative 3 and 6 months, when patients come for control, it will be learned from the patient whether they have pain, and if there is any pain, whether any procedure is applied for this pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Thoracotomy patients

Exclusion Criteria:

1. Body mass index over 35
2. A history of allergy to drugs to be used in the study
3. Chronic pain reliever use
4. Patients who refuse to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
analgesia | 48 hours
  postoperative analgesia assesment with visual analog score

SECONDARY OUTCOMES:
analgesia | 3 months
  postoperative analgesia assesment with visual analog score
analgesia | 6 months
  postoperative analgesia assesment with visual analog score

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM Y YILDIRIMGUCLU, Principal Investigator — Ankara University
Locations (1):
- Cigdem Yildirim Guclu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No